CLINICAL TRIAL: NCT04046705
Title: A Prospective Multicenter Trial Comparing Allogeneic Matched Related Haematopoietic Stem Cell Transplantation After a Reduced Intensity Conditioning Regimen, With Standard of Care in Adolescents and Adults With Severe Sickle Cell Disease
Brief Title: Comparison of Allogeneic Matched Related Haematopoietic Stem Cell Transplantation After a Reduced Intensity Conditioning Regimen With Standard of Care in Adolescents and Adults With Severe Sickle Cell Disease
Acronym: DREPA-RIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K170912J
Record Dates: First submitted 2019-07-15; First posted 2019-08-06 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLA matched haematopoietic stem cell transplantation (Experimental): Peripheral blood stem cell from matched HLA related donor.
  Interventions: Procedure: Allogeneic matched related haematopoietic stem cell transplantation
- Control arm (Other): Best standard care : Patients will receive the best standard care according to their situation and their previous treatment: initiation of Hydroxyurea, continuation or optimization of the dose of Hydroxyurea, initiation or continuation of TP, initiation of a new drug proved to improve SCD and having authorization to use in France.
  Interventions: Other: Standard arm

INTERVENTIONS:
Procedure: Allogeneic matched related haematopoietic stem cell transplantation — Allogeneic matched related haematopoietic stem cell transplantation after a reduced intensity conditioning regimen
  Arms: HLA matched haematopoietic stem cell transplantation
Other: Standard arm — In the standard arm, patients who will not be transplanted, will receive the best standard care according to their situation and their previous treatment: initiation of hydroxyurea, continuation or optimization of the dose of hydroxyurea, initiation or continuation of transfusion program, initiation of a new drug proved to improve SCD and having authorization to use in France
  Arms: Control arm

SUMMARY:
Although the survival of children with sickle cell disease (SCD) has dramatically improved over the last decades in the US and Europe, mortality remains high in adults. Moreover, many children and most adults develop a chronic debilitating condition due to organ damage. Allogeneic hematopoietic stem cell transplantation (HSCT) is currently the unique curative approach; it allows the cure of more than 95% of children transplanted from a matched related donor (MRD) after a myeloablative conditioning regimen.To date, few studies have addressed the role of HSCT in SCD adults, due to the risk of graft versus host disease (GVHD) and to the toxicity expected in older patients with a higher risk of organ damage. The development of safe, non-myeloablative conditioning regimens that allow stable mixed chimerism and avoid GVHD appears as an attractive option for HSCT to cure adults with severe SCD. The investigators design a prospective multicenter trial targeting patients over 15 years with severe SCD, and compare non-myeloablative transplant (when a matched related donor (MRD) is identified) versus no HSCT (for patients lacking MRD). The main objective is to assess the benefit of HSCT on the 2-year event free survival compared to standard care. The primary endpoint is the 2-year event free survival.

ELIGIBILITY:
Inclusion criteria

* SCD patients (SS/Sβ0)
* Aged :15 to 45 years
* With at least one non-SCD sibling > 18 years from the same parental couple
* Who presented at least one of the following criteria:
* 3 VOC requiring hospitalization over one year within the past 2 years and at least a past history of an ACS
* At least 1 ACS within the past 2 years requiring transfusions
* History of ischemic stroke or cerebral/cervical arterial stenosis > 50%
* Pulmonary hypertension defined by mean pulmonary artery pressure ≥ 25 mmHg at rest, determined by right heart catherization
* Requiring treatment with Hydroxyurea or chronic transfusion, or already treated by Hydroxyurea or transfusion program (TP) at inclusion.
* Patients already receiving chronic transfusions for VOC or ACS not responding to hydroxyurea, will be eligible, provided at least 3 VOC requiring hospitalization/year within the 2 years before initiation of chronic transfusions, and at least past history of an ACS.
* Contraception during all the study period by sirolimus for women of child bearing potential
* Signed informed consent
* Amenable to HLA typing, HSCT if an HLA-identical sibling is available.
* Patients affiliated to the French health care insurance

Exclusion Criteria

* Performance status: ECOG scale>1
* Pulmonary function: FEV1 et CVF < 50% of the theorical value
* Post capillary and severe pre-capillary pulmonary hypertension with measured mean pulmonary artery pressure at rest >35 mmHg
* Cardiac ejection fraction < 45%
* Estimated glomerular fraction rate (GFR) <50ml/mn /1.73m2
* Conjugate bilirubin >50 µmole/L, cirrhosis, ALT>4N
* Uncontrolled infection
* Known hypersensitivity of alemtuzumab
* Known hypersensitivity to murine proteins and to the following excepients: disodium edetate, polysorbate 80, potassium chloride, potassium phosphate monobasic, sodium chloride, dibasic sodium phosphate, water for injections
* Positivity for HIV
* Pregnancy or breast-feeding women
* Alloimmunization or Delayed Hemolytic Transfusion Reaction precluding red cell transfusions

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
2 year event-free survival | 2 years post-inclusion
  An event will be defined as :
  * death from any cause
  * or acute grade II-IV GVHD according to the Magic consortium 2016 classification or a moderate or severe chronic GVHD according to the NIH classification
  * or 3 hospitalizations for VOC defined according to usual criteria
  * or one ACS defined by usual clinical criteria and a pulmonary infiltrate on chest film and/or thoracic computed-tomography (CT) scan
  * or a stroke defined as a clinical event confirmed by an MRI
  * or a cerebral or cervical stenosis >25% in a new territory, or increase >25% of previous stenosis evaluated MRI and MRI
  * or a increased of at least +10% of tricuspid regurgitation velocity, (confirmed by 2 echocardiography performed with a delay of at least 3 months) compared with pre-inclusion value for patients with TRV≥2.7 at inclusion

SECONDARY OUTCOMES:
Overall survival | 2 years post-inclusion
Number of days requiring hospitalization | 1 year
  Number of days requiring hospitalization at 1 year post-inclusion with exclusion of the 5 first months post-inclusion
Number of days requiring hospitalization | 2 years post-inclusion
  Number of days requiring hospitalization at 2 years post-inclusion with exclusion of the 5 first months post-inclusion
Number of vaso-occlusive crisis (VOC) requiring hospitalization | 1 year post-inclusion
Number of vaso-occlusive crisis (VOC) requiring hospitalization | 2 years post-inclusion
Number of acute chest syndrome (ACS) requiring hospitalization | 1 year post-inclusion
Number of acute chest syndrome (ACS) requiring hospitalization | 2 years post-inclusion
Number of hospitalizations in intensive care unit | 1 year post-inclusion
Number of hospitalizations in intensive care unit | 2 years post-inclusion
Number of priapism | 1 year post-inclusion
Number of priapism | 2 years post-inclusion
Number of stroke episodes | 1 year post-inclusion
Number of stroke episodes | 2 years post-inclusion
LDH count | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in LDH
Percentage of patients with an aminotransferase value higher than five times the normal value | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in aminotransferase
Percentage of patients with a gamma-GT value higher than five times the normal value | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in gamma-GT
Percentage of patients with an Alkaline phosphatase value higher than five times the normal value | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in alkaline phosphatase
Percentage of patients with a bilirubin value higher than three times the normal value | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in bilirubin
Percentage of patients with a prothrombin value less than 70% | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in TP
Activated partial thromboplastin time higher than 1.5 times the normal value | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in TCK
Rate of hemoglobin | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in hemoglobin level
Hematocrit | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in hematocrit
Mean corpuscular volume | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in mean corpuscular volume
Hemoglobin variants | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes of percentage of hemoglobin variants
Reticulocyte count | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in percentage of reticulocyte
White blood cells count | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in white blood cells
Platelets counts | every 3 months (from inclusion to 24 months) and at Month 1, Month 2 and Month 3 in the transplant arm
  Changes in platelet counts
Microalbuminuria/creatininuria ratio | at 3 months
Microalbuminuria/creatininuria ratio | at 6 months
Microalbuminuria/creatininuria ratio | at 12 months
Microalbuminuria/creatininuria ratio | at 24 months
Ferritin level | at 3 months
Ferritin level | at 6 months
Ferritin level | at 12 months
Ferritin level | at 24 months
Transferrin saturation level | at 3 months
Percentage of transferrin saturation | at 6 months
Percentage of transferrin saturation | at 12 months
Percentage of transferrin saturation | at 24 months
LH count | at 24 months
  Gonadic function will be measured using LH
FSH count | at 24 months
  Gonadic function will be measured using FSH
Testosterone count | at 24 months
  Gonadic function will be measured using testosterone level in men
Spermogram | at 24 months
  Gonadic function will be measured using spermogram in men
Oestrogen count | at 24 months
  Gonadic function will be measured using oestrogen level in women
AMH count | at 24 months
  Gonadic function will be measured using AMH level in women
Incidence of amenorrhea | at 24 months
  Gonadic function will be measured using incidence of amenorrhea in women
Number of parity | at 24 months
Percentage of patients with a proliferative retinopathy | at 12 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Percentage of patients with a proliferative retinopathy | at 24 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Percentage of patients with a hemorrhagic retinopathy | at 12 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Percentage of patients with a hemorrhagic retinopathy | at 24 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Percentage of patients with retinal detachment | at 12 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Percentage of patients with retinal detachment | at 24 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Proportion of patients with keratitis | at 12 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Proportion of patients with keratitis | at 24 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Proportion of patients with uveitis | at 12 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Proportion of patients with uveitis | at 24 months
  Changes in retinopathy status (appearance, disappearance, improvement, aggravation)
Tricuspid regurgitant jet velocity | at 12 months
  Heart function will be assessed by a transthoracic echocardiography and using tricuspid régurgitant jet velocity
Tricuspid regurgitant jet velocity | at 24 months
  Heart function will be assessed by a transthoracic echocardiography and using tricuspid régurgitant jet velocity
Left atrial dimension | at 12 months
  Heart function will be assessed by a transthoracic echocardiography using left atrial dimension indexed to body surface
Left atrial dimension | at 24 months
  Heart function will be assessed by a transthoracic echocardiography using left atrial dimension indexed to body surface
Left ventricular dimension | at 12 months
  Heart function will be assessed by a transthoracic echocardiography using left ventricular dimension indexed to body surface
Left ventricular dimension | at 24 months
  Heart function will be assessed by a transthoracic echocardiography using left ventricular dimension indexed to body surface
Ventricular mass index value | at 12 months
  Heart function will be assessed by a transthoracic echocardiography using ventricular mass index
Ventricular mass index value | at 24 months
  Heart function will be assessed by a transthoracic echocardiography using ventricular mass index
Left ventricular ejection fraction | at 12 months
  Heart function will be assessed by a transthoracic echocardiography using left ventricular ejection fraction
Left ventricular ejection fraction | at 24 months
  Heart function will be assessed by a transthoracic echocardiography using left ventricular ejection fraction
Forced Expiratory Volume in one second (FEV) | at 12 months
  Lung function will be evaluated Forced Expiratory Volume in one second (FEV) , %
Forced Expiratory Volume in one second (FEV) | at 24 months
  Lung function will be evaluated Forced Expiratory Volume in one second (FEV) , %
DLCO | at 12 months
  Lung function will be evaluated using DLCO the diffusion capacity of carbon monoxide
DLCO | at 24 months
  Lung function will be evaluated using DLCO the diffusion capacity of carbon monoxide
Forced vital capacity | at 12 months
  Lung function will be evaluated using forced vital capacity (FVC)
Forced vital capacity | at 24 months
  Lung function will be evaluated using forced vital capacity (FVC)
6 minutes walk test | at 12 months
  Lung function will be evaluated using 6 minutes walk test
6 minutes walk test | at 24 months
  Lung function will be evaluated using 6 minutes walk test
Number of new episodes of avascular osteonecrosis | at 24 months
Number of patients for each location of new episodes of avascular osteonecrosis | at 24 months
  Location of new episodes of avascular osteonecrosis will be assessed using radiography and magnetic resonance imaging
Fractures | at 24 months
  Number of new episodes of fractures
Central nervous system function | at 12 months
  Central nervous system function will be assessed using magnetic resonance Imaging with ARM/MRI
Central nervous system function | at 24 months
  Central nervous system function will be assessed using magnetic resonance Imaging with ARM/MRI
Iron overload | at inclusion
  Iron overload will be assessed using liver and heart magnetic resonance Imaging in patients with ferritin > 1000 microg/L
Iron overload | at 12 months
  Iron overload will be assessed using liver and heart magnetic resonance Imaging in patients with ferritin > 1000 microg/L
Iron overload | at 24 months
  Iron overload will be assessed using liver and heart magnetic resonance Imaging in patients with ferritin > 1000 microg/L
Red blood cell packed transfused | at 24 months
  Number of red blood cell packed transfused from 6 months post-inclusion (pre and early post-transplant transfusion are a standard of care and may not be counted)
Number of delayed hemolytic transfusion reaction (DHTR) | at 3 months
  DHTR will be defined as associated with hemoglobinuria/dark urine in the month following transfusion +/- bone pain with increased hemolytic markers and drop in HbA or new RBC allo-Ab
Number of delayed hemolytic transfusion reaction (DHTR) | at 6 months
  DHTR will be defined as associated with hemoglobinuria/dark urine in the month following transfusion +/- bone pain with increased hemolytic markers and drop in HbA or new RBC allo-Ab
Number of delayed hemolytic transfusion reaction (DHTR) | at 12 months
  DHTR will be defined as associated with hemoglobinuria/dark urine in the month following transfusion +/- bone pain with increased hemolytic markers and drop in HbA or new RBC allo-Ab
Number of delayed hemolytic transfusion reaction (DHTR) | at 24 months
  DHTR will be defined as associated with hemoglobinuria/dark urine in the month following transfusion +/- bone pain with increased hemolytic markers and drop in HbA or new RBC allo-Ab
Proportion of patients with new RBC alloantibodies | at 3 months
  New RBC alloantibodies will be assessed using blood test
Proportion of patients with new RBC alloantibodies | at 6 months
  New RBC alloantibodies will be assessed using blood test
Proportion of patients with new RBC alloantibodies | at 12 months
  New RBC alloantibodies will be assessed using blood test
Proportion of patients with new RBC alloantibodies | at 24 months
  New RBC alloantibodies will be assessed using blood test
Percentage of patients with an oral opioid consumption | at 3 months
Percentage of patients with an oral opioid consumption | at 6 months
Percentage of patients with an oral opioid consumption | at 12 months
Percentage of patients with an oral opioid consumption | at 24 months
Quality of life evaluated using MOS SF36 questionnaire | at 3 months
  Quality of life evaluated using MOS SF36 questionnaire (Medical Outcomes Study - 36-Item Short Form Health Survey). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are grouped into three categories: functional status, well-being, overall health assessment. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). For each dimension, the scores for the different items are coded and then summed and transformed linearly on a scale ranging from 0 to 100. A physical composite score and a mental composite score can be calculated according to an established algorithm
Quality of life evaluated using MOS SF36 questionnaire | at 6 months
  Quality of life evaluated using MOS SF36 questionnaire (Medical Outcomes Study - 36-Item Short Form Health Survey). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are grouped into three categories: functional status, well-being, overall health assessment. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). For each dimension, the scores for the different items are coded and then summed and transformed linearly on a scale ranging from 0 to 100. A physical composite score and a mental composite score can be calculated according to an established algorithm
Quality of life evaluated using MOS SF36 questionnaire | at 12 months
  Quality of life evaluated using MOS SF36 questionnaire (Medical Outcomes Study - 36-Item Short Form Health Survey). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are grouped into three categories: functional status, well-being, overall health assessment. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). For each dimension, the scores for the different items are coded and then summed and transformed linearly on a scale ranging from 0 to 100. A physical composite score and a mental composite score can be calculated according to an established algorithm
Quality of life evaluated using MOS SF36 questionnaire | at 24 months
  Quality of life evaluated using MOS SF36 questionnaire (Medical Outcomes Study - 36-Item Short Form Health Survey). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are grouped into three categories: functional status, well-being, overall health assessment. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). For each dimension, the scores for the different items are coded and then summed and transformed linearly on a scale ranging from 0 to 100. A physical composite score and a mental composite score can be calculated according to an established algorithm
Depression and Anxiety status | at 3 months
  Depression and anxiety will be assessed using Hospital Anxiety and Depression Scale (HADS) questionnaire. The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Depression and Anxiety status | at 6 months
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Depression and Anxiety status | at 12 months
  Depression and anxiety will be assessed using Hospital Anxiety and Depression Scale (HADS) questionnaire. The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Weight | at 3 months
  Evolution of weight
Weight | at 6 months
  Evolution of weight
Weight | at 12 months
  Evolution of weight
Weight | at 24 months
  Evolution of weight
Number of severe infections | at 24 months
  A severe infection will be defined as a CTAE score of grade 3 or 4
GvHD incidence | at 12 months
GvHD incidence | at 24 months
Grading of GvHD | at 12 months
  Grading of GvHD will be assessed using magic consortium 2016 and NIH classification
Chimerism in HSCT | at 1 month
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletion
Chimerism in HSCT | at 2 months
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletion
Chimerism in HSCT | at 3 months
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletion
Chimerism in HSCT | at 6 months
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletionchimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant.
Chimerism in HSCT | at 9 months
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletion
Chimerism in HSCT | at 12 months
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletion
Chimerism in HSCT | at 18 months
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletion
Chimerism in HSCT | at 24 months
  Chimerism in HSCT will be assessed on total blood population and on T subset. In patients transplanted in Paris area, a more extensive centralized chimerism will be performed if donor T lymphocyte chimerism will be under 70% at 3 months post-transplant. Chimerism analysis by PCR microsatellite or by quantitative real-time PCR of insertion/deletion
Number of days of hospitalization | Number of days of hospitalization from inclusion at M24
  Number of days of hospitalization from inclusion
RBC and WBC adherence | at inclusion
  Study of RBC and WBC adherence on lymphocytes subpopulation (including NK-T cells). Modulation of WBC and RBC surface markers by allograft.
RBC and WBC adherence | at 12 months
  Study of RBC and WBC adherence on lymphocytes subpopulation (including NK-T cells). Modulation of WBC and RBC surface markers by allograft.
RBC and WBC adherence | at 24 months
  Study of RBC and WBC adherence on lymphocytes subpopulation (including NK-T cells). Modulation of WBC and RBC surface markers by allograft.
Expression of RBC and WBC surface markers | at inclusion
  Expression of RBC and WBC surface markers on lymphocytes subpopulation
Expression of RBC and WBC surface markers | at 12 months
  Expression of RBC and WBC surface markers on lymphocytes subpopulation
Expression of RBC and WBC surface markers | at 24 months
  Expression of RBC and WBC surface markers on lymphocytes subpopulation
Mast cell mediator release | at inclusion
  Master cell mediator release will be assessed using plasma sample. Modulation of mast cell mediators release by allograft (tryptase, substance P and histamine)
Mast cell mediator release | at 12 months
  Master cell mediator release will be assessed using plasma sample. Modulation of mast cell mediators release by allograft (tryptase, substance P and histamine)
Mast cell mediator release | at 24 months
  Master cell mediator release will be assessed using plasma sample. Modulation of mast cell mediators release by allograft (tryptase, substance P and histamine)
Inflammatory cytokines | at inclusion
  Inflammatory cytokines will be measured using serum sample. Modulation of inflammatory cytokine (TNF-alpha, IL-1, IL-6...) by allograft
Inflammatory cytokines | at 12 months
  Inflammatory cytokines will be measured using serum sample. Modulation of inflammatory cytokine (TNF-alpha, IL-1, IL-6...) by allograft
Inflammatory cytokines | at 24 months
  Inflammatory cytokines will be measured using serum sample. Modulation of inflammatory cytokine (TNF-alpha, IL-1, IL-6...) by allograft